CLINICAL TRIAL: NCT00459511
Title: The Importance of Adrenomedullin (AM) on Pituitary-Adrenal Axis and Glucose Kinetics in Pediatric Patients With Systemic Inflammatory Response Syndrome
Brief Title: The Importance of Adrenomedullin (AM) on ACTH-Cortisol-Glucose Axis
Acronym: AM
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Other Study IDs: FMUSP/ cappesq 675/05
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Last update posted 2007-04-12 (Estimated); Status verified 2007-04

CONDITIONS: Systemic Inflammatory Response Syndrome; Hyperglycemia
Keywords: Adrenomedullin; Glucose; Insulin; Systemic Inflammatory response Syndrome; Pediatric; Cortisol; ACTH
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome; Hyperglycemia; Insulin Resistance | interventions — Interleukin-6; Adrenocorticotropic Hormone; Hydrocortisone; Glucose; Insulin

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Blood AM, IL-6, ACTH, Cortisol, Glucose and Insulin

SUMMARY:
Hyperglycemia is frequent manifestations of the human metabolic response to systemic inflammatory response syndrome (SIRS),sepsis and septic shock, and are implicated in the clinical outcome.

Adrenomedullin is elevated in SIRS, sepsis and septic shock and has been demonstrated the inhibitory role on insulin and adrenocorticotropic hormone secretion.

Our hypothesis is that: AM elevation after SIRS could be the responsible to maintain hyperglycemia

DETAILED DESCRIPTION:
Studies in cultured vascular endothelial cells and vascular smooth muscle cells demonstrate that cytokines strongly stimulate adrenomedullin production and release.

Adrenomedullin has been measured in a wide range of clinical researches. Of all conditions investigated, the greatest increment in plasma adrenomedullin has been observed in septic shock. It appears that AM is directly responsible for the hypotension characteristic of septic shock. Studies have shown that administration of AM and AMBP-1 before the onset of sepsis (i.e., pretreatment) prevents transition from the hyperdynamic phase to the hypodynamic phase in the progression of sepsis, attenuates tissue and organ damage, and reduces sepsis-induced mortality.

Two groups described the effects of AM on the pituitary. Taken together, these studies suggest that AM has a role in inhibiting ACTH release.

Mulder et al. first reported the stimulatory effects of adrenomedullin on insulin secretion from isolated rat islets. In direct contrast to this, Martínez et al. clearly demonstrated the inhibitory role of adrenomedullin on insulin secretion in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Children above 2 years, submitted to elective cardiopulmonary bypass (CPB, only interatrial or ventricular communication) with no endocrine disease or infection.

Exclusion Criteria:

* Children with endocrine disease, undernutrition, with some medication that might interfere in the study (corticosteroids.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2006-01; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thelma Okay, PHD, Study Director — Childrens Institute / Molecular Biology
Locations (1):
- Childrens Institute, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Martinez A, Weaver C, Lopez J, Bhathena SJ, Elsasser TH, Miller MJ, Moody TW, Unsworth EJ, Cuttitta F. Regulation of insulin secretion and blood glucose metabolism by adrenomedullin. Endocrinology. 1996 Jun;137(6):2626-32. doi: 10.1210/endo.137.6.8641217.
- [Result] Zhou M, Simms HH, Wang P. Adrenomedullin and adrenomedullin binding protein-1 attenuate vascular endothelial cell apoptosis in sepsis. Ann Surg. 2004 Aug;240(2):321-30. doi: 10.1097/01.sla.0000133253.45591.5b. PMID 15273558
- [Result] Koo DJ, Zhou M, Chaudry IH, Wang P. The role of adrenomedullin in producing differential hemodynamic responses during sepsis. J Surg Res. 2001 Feb;95(2):207-18. doi: 10.1006/jsre.2000.6013. PMID 11162047
- [Result] Yoshikawa D, Kawahara F, Okano N, Hiraoka H, Kadoi Y, Fujita N, Morita T, Goto F. Increased plasma concentrations of the mature form of adrenomedullin during cardiac surgery and hepatosplanchnic hypoperfusion. Anesth Analg. 2003 Sep;97(3):663-670. doi: 10.1213/01.ANE.0000072543.78106.AA. PMID 12933380
- [Result] Takeuchi M, Morita K, Iwasaki T, Toda Y, Oe K, Taga N, Hirakawa M. Significance of adrenomedullin under cardiopulmonary bypass in children during surgery for congenital heart disease. Acta Med Okayama. 2001 Aug;55(4):245-52. doi: 10.18926/AMO/31995. PMID 11512567
- [Result] Rossi GP, Conconi MT, Malendowicz LK, Nussdorfer GG. Role of the endogenous adrenomedullin system in regulating the secretion and growth of rat adrenal cortex. Hypertens Res. 2003 Feb;26 Suppl:S85-92. doi: 10.1291/hypres.26.s85. PMID 12630816
- [Result] Kapas S, Martinez A, Cuttitta F, Hinson JP. Local production and action of adrenomedullin in the rat adrenal zona glomerulosa. J Endocrinol. 1998 Mar;156(3):477-84. doi: 10.1677/joe.0.1560477. PMID 9582504